CLINICAL TRIAL: NCT02702037
Title: Older Person's Exercise and Nutrition Study (OPEN): a Simple Physical Exercise Combined With Protein Supplement - Effects on Functional Status and Independence Among Older People: A Cluster Randomised Controlled Trial
Brief Title: Older Person's Exercise and Nutrition Study
Acronym: OPEN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Principal Investigator, Anne-Marie Bostrom, Associate Professor, Senior Lecturer, Karolinska Institutet
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: ISS.FinGrant_Fortimel_2015
Record Dates: First submitted 2016-02-26; First posted 2016-03-08 (Estimated); Last update posted 2019-04-26 (Actual); Status verified 2019-04

CONDITIONS: Mobility Limitations; Malnutrition
MeSH Terms: conditions — Mobility Limitation; Malnutrition | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The participants will be supported to perform the sit-to-stand exercise at least four times per day during 12 weeks (7 days/week).
  The participants will also be offered an oral protein-rich supplement (125 ml, 18 g protein (24% of RDI), 300 kcal) twice a day in conjunction with two of the four sit-to-stand exercises during 12 weeks (7 days/week).
  Interventions: Dietary Supplement: oral protein-rich supplement; Other: Exercise
- Control (No Intervention): Standard care

INTERVENTIONS:
Dietary Supplement: oral protein-rich supplement — The older person will be offered an oral protein-rich supplement (125 ml, 18 g protein (24% of RDI), 300 kcal) twice a day in conjunction with two of the four sit-to-stand exercises during 12 weeks (7 days/week).
  Arms: Intervention
Other: Exercise — The older person will get up from a chair to stand and then sit down again repeatedly at least four times per day, 7 days during 12 weeks
  Other Names: Sit-to-stand
  Arms: Intervention

SUMMARY:
The novelty with the OPEN study is to evaluate the effects of the simple sit-to-stand exercise during routine care, in combination with an oral protein-rich supplement, on functional status and independence in frail older persons. In this study we will also explore the experiences among older persons in the intervention group as wells as among staff of promoting the sit-to-stand exercise and nutritional supplement to gain knowledge for implementation as a daily routine in nursing homes across Sweden.

Hypothesis The main hypothesis of the OPEN study is that physical exercise performed as a daily routine along with an oral protein-rich supplement, will result in improved functional status and independence in everyday life activities and thereby enhance health-related quality of life in older persons living in nursing homes. The primary outcome measure for functional status will be the number of sit-to-stands that the participant is able to complete in 30 seconds.

Specific aims Aim I: To study the effects of the sit-to-stand exercise combined with an oral protein-rich supplement on functional and nutritional status, and health-related quality of life, and the frequency and incidence of falls, pressure ulcers and incontinence in older persons living in nursing homes. Furthermore, the cost effectiveness of the combination of the sit to stand exercise and oral protein-rich supplement vs. the control group will also be examined.

Aim II: To describe the older persons' perceptions of daily being offered to conduct the sit-to-stand exercise and to drink the nutritional supplement.

Aim III: To describe staff's perceptions of supporting the sit-to-stand exercise and the nutritional supplement with older persons living in nursing homes.

ELIGIBILITY:
Inclusion Criteria:

* Able to rise independently from a seated position to standing-

Exclusion Criteria:

* BMI >30
* severe dysphagia,
* tube feeding,
* severe kidney failure,
* bedridden people,
* terminal stage of life
* Lack of informed consent.

Min Age: 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 120 (Actual)
Dates: Start 2016-03-01 (Actual); Primary Completion 2017-12-11 (Actual); Study Completion 2017-12-11 (Actual)

PRIMARY OUTCOMES:
The primary outcome measure for functional status will be the number of sit-to-stands that the participant is able to complete in 30 seconds | 12 weeks

SECONDARY OUTCOMES:
Functional balance | 12 weeks
  Bergs Balance Scale
Walking ability | 12 weeks
  walking propulsion indoors for a distance of 10 m at self-selected speed
Everyday activities and function | 12 weeks
  Functional Independence Measure (FIM) which comprises 18 items grouped in the following functional domains: bathing, bowel management, toileting, eating, dressing lower body and social interaction. It is scored on a 7-point scale from 1 (dependent) to 7 (independent). 29. Cohen ME & Marino RJ. The tools of disability outcomes research functional status measures. Arch Phys Med Rehabil 2000;81:21-29
Nutritional status | 12 weeks
  Mini Nutritional Assessment,
Body composition | 12 weeks
  bioelectrical impedance analysis
Blood Chemistry - albumin | 12 weeks
  plasma albumin
Blood Chemistry - transthyretin | 12 weeks
  plasma transthyretin
Blood Chemistry - CRP | 12 weeks
  plasma C-reactive protein (CRP)
Blood Chemistry - IGF-1 | 12 weeks
  The anabolic mediator plasma insuline-like growth factor-1 (IGF-I)
Blood Chemistry - S-25 vit D | 12 weeks
  D-vitamin status will be assessed by S-25 (OH) vitamin D
Blood Chemistry - creatinin | 12 weeks
  Plasma creatinin
Blood Chemistry - Cystatin C | 12 weeks
  Plasma-Cystatin C
Quality of Life | 12 weeks
  EQ-5D, the Euroqool instrument
Healthcare Resource Use - hospitalisations | 12 weeks
  hospitalisations
Healthcare Resource Use - length of stay | 12 weeks
  length of stay at hospital
Healthcare Resource Use - number of visits | 12 weeks
  the number of visits to healthcare professionals (both as outpatients and as a home visit
Healthcare Resource Use - time of staff | 12 weeks
  the time of the staff (nursing aides) in the training and implementation of the intervention
Medical incidences - fall | 12 weeks
  frequency and incidence of falls
Medical incidences - pressure ulcers | 12 weeks
  frequency and incidence of pressure ulcers
Medical incidences - infections | 12 weeks
  frequency and incidence of infections
Medical incidences - incontinence | 12 weeks
  frequency and incidence of incontinence

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Marie Bostrom, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Stockholms Sjukhem, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vikstrom S, Gronstedt HK, Cederholm T, Franzen E, Faxen-Irving G, Seiger A, Bostrom AM. Experiences of supporting older persons in completion of an exercise and nutrition intervention: an interview study with nursing home staff. BMC Geriatr. 2021 Feb 5;21(1):109. doi: 10.1186/s12877-021-02039-7. PMID 33546610
- [Derived] Vikstrom S, Gronstedt HK, Cederholm T, Franzen E, Seiger A, Faxen-Irving G, Bostrom AM. A health concept with a social potential: an interview study with nursing home residents. BMC Geriatr. 2020 Sep 4;20(1):324. doi: 10.1186/s12877-020-01731-4. PMID 32887570
- [Derived] Gronstedt H, Vikstrom S, Cederholm T, Franzen E, Luiking YC, Seiger A, Wimo A, Faxen-Irving G, Bostrom AM. Effect of Sit-to-Stand Exercises Combined With Protein-Rich Oral Supplementation in Older Persons: The Older Person's Exercise and Nutrition Study. J Am Med Dir Assoc. 2020 Sep;21(9):1229-1237. doi: 10.1016/j.jamda.2020.03.030. Epub 2020 May 26. PMID 32471657
- [Derived] Gronstedt H, Vikstrom S, Cederholm T, Franzen E, Seiger A, Wimo A, Faxen-Irving G, Bostrom AM. A study protocol of Older Person's Exercise and Nutrition Study (OPEN) - a sit-to-stand activity combined with oral protein supplement - effects on physical function and independence: a cluster randomized clinical trial. BMC Geriatr. 2018 Jun 7;18(1):138. doi: 10.1186/s12877-018-0824-1. PMID 29898671